CLINICAL TRIAL: NCT05431517
Title: Incidence, Risk Factors and Endoscopic Retrieval of Proximally Migrated Pancreatic Stents: 25 Years of Experience in a Tertiary Center
Brief Title: Incidence, Risk Factors and Endoscopic Retrieval of Proximally Migrated Pancreatic Stents
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Professor, Changhai Hospital
Other Study IDs: IREPS20220611
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Stenting; Pancreatic Stent Displacement
Keywords: Endoscopic retrograde cholangiopancreatography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-migration group: Cases without migration after pancreatic stenting under ERCP.
  Interventions: Procedure: Analysis of ERCP records
- Migration group: Cases with migration after pancreatic stenting under ERCP.
  Interventions: Procedure: Analysis of ERCP records

INTERVENTIONS:
Procedure: Analysis of ERCP records — Data will be extracted from ERCP records of stenting, mainly including: 1) Age at the time of ERCP; 2) Gender; 3) Indication; 4) Papilla selection (major or minor); 5) Whether endoscopic sphincterotomy (EST) was performed; 6) Presence of nipple diverticulum; 7) Morphology of the pancreatic duct; 8) Status of pancreatic duct stones; 9) Number, shape, material, diameter and length of the stent; and 10) Operation of the bile duct. Additional data were extracted from the pertinent ERCP records of stent migration: 1) Shape, material, diameter and length of the displaced stent; 2) Type of migration; and 3) Removal tools.

SUMMARY:
This study intends to determine the incidence, risk factors and endoscopic treatment of proximally migrated pancreatic stents.

DETAILED DESCRIPTION:
Endoscopic pancreatic stenting can be used to treat a variety of pancreatic disorders, including chronic pancreatitis-induced pancreatic duct stenosis, pancreatic schizophrenia, pancreatic leakage, pancreatic pseudocyst drainage, and prophylactic pancreatic duct stenting. Postoperative stent migration is one of the complications associated with pancreatic stent placement.

In this retrospective study, more than 9,000 Endoscopic retrograde cholangiopancreatography (ERCP) cases at our center over the past 25 years will be analyzed to determine the incidence, risk factors and endoscopic treatment of proximally migrated pancreatic stents.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic stent placement under ERCP;
* Pancreatic stent migration found by ERCP;
* Displaced pancreatic stent removal by ERCP technique.

Exclusion Criteria:

* Incomplete ERCP records (e.g., missing stent size information);
* Immediate removal of pancreatic stent following implantation for a variety of reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with placements of pancreatic stents under ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 9073 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence of proximally migrated pancreatic stents | Within 1 month after data analysis
Success rate of endoscopic removal of migrated pancreatic stents | Within 1 month after data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Liang-hao Hu, MD, Principal Investigator — Changhai Hospital
Locations (1):
- Changhai Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No